CLINICAL TRIAL: NCT00740103
Title: Long-term Study of Semapimod (CNI-1493) for Treatment of Moderate to Severe Crohn's Disease With Reference to Study CNI-1493-CD-04, 1 or 3 Days' Treatment vs. Placebo
Brief Title: Long-term Study of Semapimod (CNI-1493) for Treatment of Crohn's Disease
Acronym: CD05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNI-1493-CD05
Record Dates: First submitted 2008-08-21; First posted 2008-08-22 (Estimated); Last update posted 2025-03-28 (Actual); Status verified 2012-08

CONDITIONS: Crohn's Disease
Keywords: Semapimod; Crohn's Disease; TNF-alpha inhibitor; MAP Kinase inhibitor; CNI-1493
MeSH Terms: conditions — Crohn Disease | interventions — semapimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Semapimod 60 mg IV x 3 days q 6 - 8 weeks
  Interventions: Drug: Semapimod

INTERVENTIONS:
Drug: Semapimod — 60 mg IV x 3 days q 6 - 8 weeks
  Other Names: CNI-1493

SUMMARY:
CNI-1493-CD05 is an open-label extension study of CNI-1493-CD04. In the CD05 study, patients are eligible for up to 5 courses of semapimod 60 mg IV x 3 days every 6 - 8 weeks. Primary objective is assessment of the efficacy of cumulative doses of semapimod measured by decrease in Crohn's Disease Activity Index (CDAI).

DETAILED DESCRIPTION:
CNI-1493-CD05 is an open-label extension study of CNI-1493-CD04. In the CD05 study, patients are eligible for up to 5 courses of semapimod 60 mg IV x 3 days every 6 - 8 weeks. Primary objective is assessment of the efficacy of cumulative doses of semapimod measured by decrease in Crohn's Disease Activity Index (CDAI). In addition, the safety of repeated courses was measured by recording adverse events over time.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria

1. Patients satisfactorily completing study CNI-1493-04 were eligible for participation in this study. Satisfactory completion was defined as follows:

   1. The patient met all eligibility criteria for participation in study CNI-1493-04 or was granted an exemption by the medical monitor for factors indicating ineligibility.
   2. The patient received at least 2 of the 3 planned doses of study medication.
   3. The patient had no adverse event >grade 2 felt to be possibly, probably or definitely related to study medication.
   4. The patient underwent all required evaluations, both for safety and efficacy, at baseline and day 29 and, for patients enrolling between days 43 and 57 of study CNI-1493-CD-04, at least one full later evaluation, ie the procedures required at day 43 and/or 57.
2. At baseline for study CNI-1493-CD-05, patients were to meet the same concomitant medication criteria as for study CNI-1493-CD-04:

   1. Patients receiving medications for CD were to be on each medication for at least 8 weeks prior to screening and on stable doses of each for at least 2 weeks prior to baseline assessments, with the following exceptions:

      * those on methotrexate were to be on a stable dose for at least 4 weeks and must not be receiving more the 25mg/week
      * those on azathioprine or 6-mercaptopurine on a stable dose for at least 10 weeks
      * those on corticosteroids were to have been on them for at least 2 weeks and on a stable for those 2 weeks. They were not to be receiving more than 20 mg/day prednisone (or equivalent).
      * those on mesalazine were to have been on for at least 6 weeks and on a stable dose for at least 2 weeks
      * those on antibiotics for CD were to have been on for at least 2 weeks and on a stable dose for those 2 weeks
   2. Patients who were not using other CD medications were to have stopped any previous use of these agents at least 4 weeks prior to baseline assessment for study CNI-1493-CD-05.
3. Patients were required to sign informed consent specifically for this study, in addition to the consent for study CNI-1493-CD-04.
4. Men and women of childbearing potential were to be using a barrier method (diaphragm or condom) of contraception and continue doing so for at least 3 months after last study medication. It was strongly recommended that two forms be used.
5. Patients were to be able to adhere to the study visit schedule and/or protocol requirements.

Exclusion Criteria:

Only patients completing CD04 were eligible and must not have met any of the exclusion criteria for that study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2002-12; Primary Completion 2004-07 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Crohn's disease activity index (CDAI) | Every 6 - 8 weeks

SECONDARY OUTCOMES:
Safety measured by adverse events | Every 6 - 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daan Hommes, MD, Principal Investigator — Academic Medical Center, Netherlands
Locations (26):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Advanced Gastroenterology Associates, Suwanee, Georgia
  - Northwestern University, Chicago, Illinois
  - Long Island Clinical Research Associates, Great Neck, New York
  - Asher Kornbluth, MD, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Gastroenterology Associates, Bristol, Tennessee
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Academic Hospital Gasthuisberg, Leuven
- Germany (7):
  - Benjamin Franklin University, Berlin
  - Medizinischen Hochschule-Hannover, Hanover
  - Universitats Klinikum Heidelberg, Heidelberg
  - University of Kiel, Kiel
  - Gastroenterologische Fachpraxis, Minden
  - Stadtisches Krankenhaus Munchen-Bogenhausen, München
  - University of Munster, Münster
- Israel (5):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Hospital, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - Free University (Vrije Universiteit), Amsterdam
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Erasmus Medical Center, Rotterdam